CLINICAL TRIAL: NCT00487058
Title: A Phase I Dose Escalation Study of LBQ707 (Gimatecan) Administered Orally Twice Per Week to Japanese Patients With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBQ707A1103
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Advanced Solid Tumors
Keywords: Gimatecan; topoisomerase I inhibitor; advanced solid tumors
MeSH Terms: interventions — ST 1481

INTERVENTIONS:
Drug: Gimatecan

SUMMARY:
This study assesses the tolerability, safety, efficacy and pharmacokinetics of gimatecan in Japanese patients. Gimatecan is administered orally twice per week, every 28 days, to adult patients with advanced solid tumors who have progressed despite standard therapy or for whom standard systemic therapy dose not exist.

ELIGIBILITY:
Inclusion criteria

* Patients with histological or cytological confirmed advanced solid tumors, which progressed despite standard therapy or for whom no standard therapy exists
* Life expectancy of at least 3 months
* No dysfunction of bone marrow
* No major impairment of renal and hepatic function

Exclusion criteria

* Gastrointestinal dysfunction, such as gastrectomy or malabsorption syndrome, that could alter absorption of the study drug
* Receipt of any investigational compound within the 28 days prior to the first dose of study drug, or failure to recover from the side effects of such prior therapy
* Receipt of other antineoplastic therapy including chemotherapy, hormone therapy, immunotherapy, radiation therapy within the 28 days
* Patients known to be HIV, or hepatitis B or C viruses positive, or patients with the presence of active or suspected acute or chronic uncontrolled infection
* Patients with a history of allergies to the camptothecin family of drugs

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by Adverse Events Characterization of the pharmacokinetic profile of gimatecan Anti-tumor activity assessed by Response Evaluation Criteria in Solid Tumors RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Saitama Prefecture, Japan